CLINICAL TRIAL: NCT02219503
Title: An Open-Label, Single-Arm Study to Evaluate the Safety and Efficacy of Ombitasvir/ABT-450/Ritonavir and Dasabuvir in Adults With Genotype 1b Chronic Hepatitis C Virus (HCV) Infection and Cirrhosis (TURQUOISE-III)
Brief Title: A Study to Evaluate the Safety and Efficacy of Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir in Adults With Genotype 1b Chronic Hepatitis C Virus (HCV) Infection and Cirrhosis
Acronym: TURQUOISE-III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-490; 2014-001953-18 (EudraCT Number)
Record Dates: First submitted 2014-08-15; First posted 2014-08-19 (Estimated); Results first posted 2016-06-29 (Estimated); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Chronic Hepatitis C Infection; Compensated Cirrhosis
Keywords: Hepatitis C; Chronic Hepatitis C; Compensated Cirrhosis; Cirrhotic; Hepatitis C Genotype 1b; Hepatitis C Virus; Interferon-Free; Child Pugh A; Ribavirin-Free
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — ombitasvir; paritaprevir; Ritonavir; dasabuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ombitasvir/Paritaprevir/Ritonavir plus Dasabuvir (Experimental): Ombitasvir/Paritaprevir/Ritonavir (25/150/100 mg once daily) and Dasabuvir (250 mg twice daily) administered for 12 weeks
  Interventions: Drug: Ombitasvir/Paritaprevir/Ritonavir; Drug: Dasabuvir

INTERVENTIONS:
Drug: Ombitasvir/Paritaprevir/Ritonavir — Tablet; paritaprevir co-formulated with ritonavir and ombitasvir
  Other Names: ABT-267 also known as ombitasvir; ABT-450 also known as paritaprevir; Ritonavir also known as norvir
Drug: Dasabuvir — Tablet
  Other Names: ABT-333

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of ombitasvir/ paritaprevir/ ritonavir and dasabuvir in adults with genotype 1b chronic hepatitis C virus (HCV) infection and cirrhosis.

DETAILED DESCRIPTION:
This was a multicenter study evaluating the efficacy and safety of ombitasvir/ paritaprevir/ritonavir and dasabuvir administered for 12 weeks in HCV genotype 1b (GT1b)-infected, treatment-naïve and previous pegylated interferon (pegIFN)/ ribavirin (RBV) treatment-experienced adults with compensated cirrhosis. The duration of the study was up to 36 weeks (not including a screening period of up to 42 days) and consisted of a 12-week Treatment Period and a 24-week Post-Treatment Period for all participants who received study drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic HCV genotype 1-infection prior to study enrollment. Chronic HCV-infection is defined as the following:

   * Positive for anti-HCV antibody (Ab) or HCV RNA > 1,000 IU/mL at least 6 months before Screening, and positive for HCV RNA and anti-HCV Ab at the time of Screening; or
   * HCV RNA > 1,000 IU/mL at the time of Screening with a liver biopsy consistent with chronic HCV-infection (or a liver biopsy performed prior to enrollment with evidence of chronic hepatitis C disease).
2. Screening laboratory result indicating HCV genotype 1b-infection.
3. Compensated cirrhosis defined as a Child-Pugh Score of 5 or 6 at Screening.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding.
2. Positive test result for Hepatitis B surface antigen (HBsAg) or positive human immunodeficiency virus (HIV) antibody (confirmed by Western Blot).
3. Any current or past clinical evidence of Child-Pugh B or C classification or clinical history of liver decompensation such as ascites (noted on physical exam), variceal bleeding, or hepatic encephalopathy.
4. Confirmed presence of hepatocellular carcinoma indicated on imaging techniques such as computed tomography (CT) scan or magnetic resonance imaging (MRI) within 3 months prior to Screening or on an ultrasound performed at Screening (a positive ultrasound result will be confirmed with CT scan or MRI.)
5. Use of contraindicated medications within 2 weeks of dosing
6. Screening laboratory analyses showing any of the following abnormal laboratory results:

   * Calculated creatinine clearance (using Cockcroft-Gault method) < 30 mL/min
   * Albumin < 2.8 g/dL
   * International normalized ratio (INR) > 1.8. Participants with a known inherited blood disorder and INR > 1.8 may be enrolled with permission of the AbbVie Study Designated Physician.
   * Hemoglobin < 10 g/dL
   * Platelets < 25,000 cells per mm3
   * Total bilirubin > 3.0 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Trinh, MD, Study Director — AbbVie

REFERENCES:
- [Background] Feld JJ, Moreno C, Trinh R, Tam E, Bourgeois S, Horsmans Y, Elkhashab M, Bernstein DE, Younes Z, Reindollar RW, Larsen L, Fu B, Howieson K, Polepally AR, Pangerl A, Shulman NS, Poordad F. Sustained virologic response of 100% in HCV genotype 1b patients with cirrhosis receiving ombitasvir/paritaprevir/r and dasabuvir for 12weeks. J Hepatol. 2016 Feb;64(2):301-307. doi: 10.1016/j.jhep.2015.10.005. Epub 2015 Oct 22. PMID 26476290
- See also: Related Info — http://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 60 subjects were enrolled and all the subjects completed the study. All 60 subjects were analyzed for both efficacy (included all participants who received at least 1 dose of study drug (ITT)) and safety.
Period: Overall Study
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir Plus Dasabuvir
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline analyses included all participants.
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir Plus Dasabuvir
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 37
Interleukin 28B (IL28B) Genotype [Number; unit: participants]
  CC | 10
  CT | 36
  TT | 14
  Missing | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks (SVR12) Post-treatment
Description: Sustained Virologic Response 12 (SVR12) is defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) less than the lower limit of quantification (< LLOQ; < 25 IU/mL) 12 weeks after the last dose of study drug.
  The primary efficacy endpoints were non-inferiority and superiority of the percentage of participants who achieved sustained virologic response 12 weeks after treatment in each treatment arm compared with the historical threshold for sofosbuvir and peginterferon (pegIFN)/RBV for the treatment of subjects with HCV GT1b infection and cirrhosis.
Time Frame: Post-treatment Day 1 to Post-treatment Week 12
Population: Efficacy analyses included all participants who received at least 1 dose of study drug (ITT).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir Plus Dasabuvir
Number analyzed (Participants) | 60
percentage of participants | 100 [94.0 to 100.0]
Statistical Analysis 1: Comparison: Ombitasvir/Paritaprevir/Ritonavir Plus Dasabuvir; Test type: Non-Inferiority or Equivalence — The non-inferiority of the Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir regimen in SVR12 to a historical threshold for sofosbuvir plus pegIFN/ ribavirin (RBV) for the treatment of participants with HCV Genotype 1b (GT1b) infection and cirrhosis was calculated using a 2-sided 95% CI from Wilson's score method. Non-inferiority was to be declared if the lower confidence bound was greater than 72.7%; Percentage of Participants = 100, 95% CI 2-sided [94.0 to 100.0] — 95% confidence interval (CI) was calculated using Wilson score method
Statistical Analysis 2: Comparison: Ombitasvir/Paritaprevir/Ritonavir Plus Dasabuvir; The superiority of the Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir regimen in SVR12 to a historical threshold for sofosbuvir plus pegIFN/ ribavirin (RBV) for the treatment of participants with HCV Genotype 1b (GT1b) infection and cirrhosis was calculated using a 2-sided 95% CI from Wilson's score method. Superiority was declared if the lower confidence bound was greater than 83.2%; Test type: Superiority or Other; Percentage of Participants = 100, 95% CI 2-sided [94.0 to 100.0] — 95% confidence interval (CI) was calculated using Wilson score method

2. Secondary Outcome: Percentage of Participants With On-Treatment Virologic Failure
Description: On-Treatment Virologic Failure is defined as confirmed HCV RNA >= LLOQ after HCV RNA < LLOQ during treatment, or confirmed increase from nadir (local minimum value) in HCV RNA [2 consecutive HCV RNA measurements > 1 log10 IU/mL above nadir] at any time point during treatment, or failure to suppress during treatment [all on-treatment values of HCV RNA >= LLOQ] with at least 6 weeks [defined as active study drug duration ≥ 36 days] of treatment.
Time Frame: Day 1 through Week 12
Population: Efficacy analyses included all participants who received at least 1 dose of study drug (ITT).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir Plus Dasabuvir
Number analyzed (Participants) | 60
percentage of participants | 0 [0.0 to 6.0]

3. Secondary Outcome: Percentage of Participants With Post-Treatment Relapse
Description: Post- Treatment Relapse is defined as confirmed HCV RNA >= LLOQ between end of treatment and 12 weeks after last actual dose of active study drug [up to and including the SVR12 assessment time point] for a participant with HCV RNA < LLOQ at Final Treatment Visit who completes treatment.
Time Frame: Post-treatment Day 1 to Post-treatment Week 12
Population: Efficacy analyses included all participants who received at least 1 dose of study drug (ITT).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir Plus Dasabuvir
Number analyzed (Participants) | 60
percentage of participants | 0 [0.0 to 6.0]

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the time of study drug administration to 30 days after last dose of study drug (12 weeks); SAEs were also collected from the time that informed consent was obtained until the end of the study (up to 42 weeks).
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir Plus Dasabuvir
Serious Adverse Events (participants affected / at risk) | 1/60
Other Adverse Events (participants affected / at risk) | 39/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ombitasvir/Paritaprevir/Ritonavir Plus Dasabuvir (N=60)
SYNCOPE (Nervous system disorders) | 1
HYPOTENSION (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ombitasvir/Paritaprevir/Ritonavir Plus Dasabuvir (N=60)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3
DIARRHOEA (Gastrointestinal disorders) | 12
DYSPEPSIA (Gastrointestinal disorders) | 4
NAUSEA (Gastrointestinal disorders) | 4
FATIGUE (General disorders) | 13
INFLUENZA (Infections and infestations) | 4
NASOPHARYNGITIS (Infections and infestations) | 4
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6
MYALGIA (Musculoskeletal and connective tissue disorders) | 4
DIZZINESS (Nervous system disorders) | 6
HEADACHE (Nervous system disorders) | 11
INSOMNIA (Psychiatric disorders) | 6
COUGH (Respiratory, thoracic and mediastinal disorders) | 4
PRURITUS (Skin and subcutaneous tissue disorders) | 6
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 3
HYPERTENSION (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.